CLINICAL TRIAL: NCT06630221
Title: A Phase II Study of Eltrombopag as a Novel Therapeutic Approach for Patients With Low-risk Myelodysplastic Syndromes (MDS) and Chronic Myelomonocytic Leukemia (CMML) With TET2 Mutations
Brief Title: Eltrombopag as a Novel Therapeutic Approach for Low-risk MDS and CMML With TET2 Mutations
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Abhay Singh, MD MPH (Other)
Responsible Party: Sponsor-Investigator, Abhay Singh, MD MPH, Principal Investigator, Case Comprehensive Cancer Center
Organization: Case Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE2924
Record Dates: First submitted 2024-10-04; First posted 2024-10-08 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Myelodysplastic Syndromes; Chronic Myelomonocytic Leukemia
Keywords: MDS; CMML
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myelomonocytic, Chronic | interventions — eltrombopag

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Eltrombopag (EPAG) (Experimental): Enrolled participants will receive EPAG 50 mg daily, 2h prior to or after meals for 1 cycle
  Interventions: Drug: Eltrombopag (EPAG)

INTERVENTIONS:
Drug: Eltrombopag (EPAG) — 50 mg, 28-day cycles, 3 initial cycles + 12 cycles on extension arm (maximum of 15 cycles)
  Other Names: Promacta

SUMMARY:
The purpose of this study is to evaluate if a study drug called eltrombopag can improve the blood cell counts in patients with low-risk Myelodysplastic Syndromes (MDS) and Chronic Myelomonocytic Leukemia (CMML) with mutations in TET2 gene, observe changes in the TET2 gene over time, and evaluate the effectiveness of the treatment. TET2 gene is one of the most frequently mutated genes (altered parts of the DNA) in MDS and CMML.

Eltrombopag is a Food and Drug Administration (FDA) approved drug for the treatment of severe aplastic anemia and low levels of platelets in patients with persistent or chronic immune thrombocytopenia (ITP) and chronic hepatitis C. Eltrombopag is considered investigational (experimental) in this study because the FDA has not approved its use in the treatment of low-risk MDS or CMML. Eltrombopag is a drug that helps stimulate the body's process of making more platelets (small components of blood that help with clotting) by interacting with specific parts of cells. This interaction starts a series of signals that encourage the growth and development of the cells that produce platelets. It was found that this drug could stop the growth of TET2 mutated cells.

DETAILED DESCRIPTION:
Epigenetic changes such as alterations in DNA methylation and histone modification play an important role in the pathophysiology of myelodysplastic syndromes (MDS). With the development of next-generation sequencing (NGS) platforms, it has become possible to identify genomic aberrations involved in the MDS epigenetics. Additionally, with the advances in therapeutic methods in MDS, several novel genomic aberrations have been reported to predict the effectiveness of specific treatment. It is becoming clear that genomic aberrations may offer more precise cancer phenotypes and help predict precise therapies for MDS patients (e.g. IDH1 and IDH2 inhibitors). TET2 gene is a member of the DNA methylation machinery and one of the most frequently mutated genes in MDS and chronic myelomonocytic leukemia (CMML; a disease entity similar to MDS with similar bone marrow dysplasia and accompanying cytopenias). TET DNA dioxygenases hydroxylate 5-methylcytosine (5mC) to 5-hydroxy-mC (5hmC), a process that leads to passive demethylation and thereby initiation of differentiation programs of hematopoietic stem cells (HSCs). TET2 mutations (TET2MT) often act as founder lesions for clonal hematopoiesis of indeterminate potential (CHIP). Our group has demonstrated that mutational exclusivity of TET2 and isocitrate dehydrogenases 1 and 2 (IDH1/2) result from production of a neomorphic natural TET2 inhibitor α-hydroxyglutarate (2HG). 2HG is selectively and synthetically lethal to TET2-deficient HSCs reliant for their survival on minimal residual dioxygenase activity supplied by less abundant TET1 and TET3. This observation inspired the idea of generating TET inhibitors as drugs selective for TET2 mutant (TET2MT) leukemia cells. Based on the structure of 2HG, investigator generated a more potent TETi76, and showed that this drug is indeed synthetically lethal to TET2MT and TET2 proficient cells. In search for alternative agents with suitable activity, investigator next performed a high throughput drug screen using an in vitro DNA dioxygenase assay. Among several hits, eltrombopag (EPAG) was unique, as it is already used in clinical practice as a thrombopoietin receptor (TPOR) agonist. Investigator showed that this agent inhibited growth of TET2MT cells in murine TET2MT models independent of its TPOR activity, and have determined its binding site and mode of action on TET dioxygenases.1 Since EPAG is an FDA approved drug with known toxicities and good tolerability, repurposing this agent as a TET inhibitor would greatly shorten the development time and thus rapidly provide a selective and well-tolerated drug for the therapy of patients with TET2MT MDS. Investigators have obtained granular molecular and response data from historical trials of EPAG/5Azacytidine in unselected MDS and aplastic anemia (AA) and were able to retrospectively assert that indeed those with TET2MT disease responded to EPAG therapy, resulting in decreased TET2MT clonal burden.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years at the time of signing the informed consent form.
* Willing and able to adhere to the study visit schedule and other protocol requirements.
* Established diagnosis of very low-, low-, or intermediate-risk MDS (IPSS-R < 3.5) and < 5% myeloblasts or CMML 0 (CMML-0, for cases with < 2% blasts in PB and < 5% blasts in bone marrow (BM)z,[14] with any one of the notable cytopenias as defined below:

  1. Hgb < 10 g/dL prior to enrollment
  2. ANC < 1.5×10^9/L
  3. Platelets < 100×10^9/L
* Must be relapsed, refractory/resistant, intolerant, or have inadequate response to therapies with known clinical benefits for MDS, such as EPOs, luspatercept, and HMAs (i.e., azacytidine or decitabine). Patients with del (5q) must have failed prior lenalidomide therapy.
* TET2 mutation performed at a frequency of at least > 5%.
* ECOG performance status of 0-2.
* Adequate organ function, defined as:

  1. Serum total bilirubin < 2x ULN, unless the subject has Gilbert's syndrome. Higher levels are acceptable if these can be attributed to ineffective erythropoiesis. In these cases, approval from the study PI is required.
  2. Creatinine clearance greater than 30 mL/min based on the Cockroft-Gault glomerular filtration rate estimation.
  3. Participants being enrolled on study on the basis of anemia, will only be eligible if folate, B12, serum iron, serum ferritin, total iron binding capacity, haptoglobin and peripheral smear within normal limits
  4. Hepatitis panel negative for Hep B and Hep C infection
  5. Negative for HIV infection
* Women of childbearing potential (WOCBP) may participate provided they have a negative serum pregnancy test at screening and a negative serum or urine pregnancy test within 72 h of starting treatment.
* WOCBP and males with partners who are WOCBP must agree to abstain from sexual intercourse or use effective contraception (methods that result in < 1% pregnancy rates) during eltrombopag therapy and for at least 7 days after the last eltrombopag dose. Males with partners who are WOCBP must agree to use a barrier method.

Exclusion Criteria:

* High- and Very High-risk MDS (per IPSS-R)
* CMML 1-2
* Prior HMA exposure
* Platelet count > 200×10^9/uL or leukocytosis of at least 25×10⁹/L
* Marrow fibrosis (any grade)
* Results of bone marrow biopsy within 1 month of study entry (screening bone marrow biopsy) indicating high-risk MDS or CMML-2.
* Elevated LFTs (aminotransferases and bilirubin) > 2x ULN
* Pre-existing cardiovascular disease (e.g., known coronary artery disease with percutaneous intervention or stroke within the last year) or arrhythmia (e.g., atrial fibrillation) associated with an increased risk of thromboembolic events, unless deemed acceptable by the enrolling treating physician.
* History of arterial or venous thromboembolism, and on anticoagulation.
* Severe hepatic impairment (Child-Pugh Class C)
* Recent history of cancer (i.e., within the past 5 years) with > 50% chance of cancer recurrence in the next 5 years
* Current or prior history of hematologic malignancy
* Known dysphagia, short-gut syndrome, gastroparesis, or other conditions that limit the ingestion or gastrointestinal absorption of drugs administered orally.
* Active uncontrolled systemic fungal, bacterial, or viral infection (defined as ongoing signs/symptoms related to the infection without improvement despite appropriate antibiotics, antiviral therapy, and/or other treatment.)
* Positive direct Coombs test
* Evidence of hypersplenism on physical exam
* Pregnant or lactating (women)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-06-17 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
Response Rate as assessed by hematologic response | At end of treatment (approximately up to 12 weeks)
  Response rate will be assessed to determine whether treatment with EPAG can induce a hematologic response. The different types of hematologic improvement are Erythroid response (non-transfusion dependent, Erythroid response (transfusion dependent), Platelet response (pretreatment, > 20 × 109/L), Platelet response (pretreatment, < 20 × 109/L), Neutrophil response, and Progression or relapse after HI (after reaching maximum dose, and on maximum dose for 12 weeks).

SECONDARY OUTCOMES:
AML-free survival | At end of treatment (approximately up to 12 weeks)
  AML-free survival will be calculated using the Kaplan-Meier method
Progression Free Survival | At end of treatment (approximately up to 12 weeks)
  Progression free survival will be calculated using the Kaplan-Meier method
Change in TET2 mutation burden as measured by variant allele fraction. | Baseline, end of cycle 3(28 days per cycle), end of treatment(approximately up to 12 weeks)
  Change in mutant TET2 variant allele fraction
Rates of robust response as measured by platelet count | Approximately at 24 weeks post administration of intervention
  Robust response will be summarized with a frequency and 95% confidence interval.
Rates of robust response as measured by hemoglobin | Approximately at 24 weeks post administration of intervention
  Robust response will be summarized with a frequency and 95% confidence interval.
Rates of robust response as measured by ANC | Approximately at 24 weeks post administration of intervention
  Robust response will be summarized with a frequency and 95% confidence interval.

CONTACTS AND LOCATIONS:
Overall Officials: Abhay Singh, MD, MPH, Principal Investigator — Case Comprehensive Cancer Center, Cleveland Clinic Taussig Cancer Institute
Locations (1):
- Case Comprehensive Cancer Center, Cleveland Clinic Foundation Taussig Cancer Institute, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in publication will be shared as a combined summary. Any individual outcomes published per subject will be de- identified utilizing the subject ID (e.g., dosing, demographics, adverse events, etc.)
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data included in the peer reviewed publication will be publicly available starting 6 months after publication and will be available indefinitely. No raw data will be shared.
Access Criteria: A peer-reviewed publication will be made available according to the publishing journal's specifications. CCF personnel will not share study data apart from that which has been published publicly.
URL: https://pubmed.ncbi.nlm.nih.gov/